CLINICAL TRIAL: NCT03079804
Title: Comparison Between Two Mobilization Techniques With and Without Ankle Thrust on Balance in Patients With Chronic Ankle Instability
Brief Title: Comparison Between Two Mobilization Techniques of Ankle on Balance in Patients With Chronic Ankle Instability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Ceara (Other)
Responsible Party: Principal Investigator, Pedro Olavo de Paula Lima, Head of Department of Physical Therapy, Universidade Federal do Ceara
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: POdePLima
Record Dates: First submitted 2017-03-06; First posted 2017-03-14 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Ankle Sprains
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Opaque envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental MWM (Experimental): Other names:
  4 mobilizations - 10 seconds 20 seconds of rest
  Interventions: Other: Experimental MWM; Other: Experimental Thrust; Other: Placebo
- Experimental Thrust (Active Comparator): Other names:
  1 traction with caudal direction in high speed and low amplitude increasing dorsiflexion.
  Interventions: Other: Experimental MWM; Other: Experimental Thrust; Other: Placebo
- Placebo (Placebo Comparator): Other names:
  It will accurately reproduce the positioning of the hand in the specific treatment condition (Thrust or MWM), however, without applying any movement or force. All interactions, procedures and deadlines will be identical.
  Interventions: Other: Experimental MWM; Other: Experimental Thrust; Other: Placebo

INTERVENTIONS:
Other: Experimental MWM — Mobilization with Movement
Other: Experimental Thrust — Mobilization grade 5 (Thrust)
Other: Placebo — Procedures similar to Experimental MWM group, but without aplly any force

SUMMARY:
The ankle joint is often affected by injuries, especially lateral sprains, often leading to chronic instability. Joint mobilization techniques seem to influence the sense of joint positioning. The objective of the study is to compare mobilization techniques in the balance of athletes with chronic ankle instability. A randomized clinical trial with participants allocated in three groups: Talocrural manipulation, mobilization with movement and placebo will be assessed in their primary endpoints and secondary balance and dorsiflexion range of motion respectively.

DETAILED DESCRIPTION:
Biodex Balance System: The unipodal stability protocol was used in the anteroposterior and laterolateral directions. The test lasts for 20 seconds with five levels of instability, with level six being more stable and level two more unstable. The participant performed an adaptation test with the system and subsequently assessed the performance of the balance in three tests in each limb between each 10-second test. This will be instructed about the positioning during its evaluation, being oriented to keep the gaze in the previous direction; Hands on waist; Contralateral knee flexed at 90º, foot positioning is referenced in degrees on the platform as anthropometric information provided on the participant. At the end, the results of the anteroposterior and lateral-lateral directions and the general index were collected.

Weight Bearing Lunge Test (WBLT): The WBLT consisting of the use of a tape measure has no soil in which the participant will support or be evaluated so that the first finger touches On the tape and its distance to a reference wall for tape measurement. Required that the participant performs ankle dorsiflexion in CCF with the purpose of approaching the knee in the wall avoiding to remove the heel of the ground, that is on a marking.

Y test: To evaluate the dynamic balance and reach of lower limbs will be used The test balance consisting of the evaluation of the participant's performance during the movements of anterior, posteromedial and posterolateral angle with the value measured in centimeters with metric tapes In Direction.

The protocol performed six replicates for adaptation and one final repeat that is considered as a result of the test. For an earlier point, the reference point used is not support for a fixed reference point for the intersection of the conditions and for two other directions used. It is necessary that the participant be the same as the member farthest from the starting point without touching the tape. At the end of the seventh repetition is measured or value and considered the test result.

Intervention: Participants are divided into three groups: Thrust Group in open kinetic chain; MWM group in closed kinetic chain and control group with placebo intervention. Allocation in one of the groups will be randomized by lot.

Taken as applications of the questionnaires and initial evaluations (BBS, WBLT, Y Test), the assays receive a specific technique, are reassessed with the BBS and WBLT.

Talocrural manipulation: The technique of talocrural manipulation consists in the application of traction with a high caudal direction. Follow with the participant in supine position and as two hands to therapist around the talocrural joint, fifth finger in the anterior talar region and the two thumbs in the plantar area do the participant performing a manipulation in the affected limb. It is not considered an audible cavitation presence.

Mobilization with Motion (MWM): The Mulligan® concept-mobilized manual therapy technique follows the following protocol: the athlete is positioned on a stretcher with the limb treated in hip and knee flexion and the contralateral limb in knee flexion And neutral hip. With the use of a belt in the hip region of the physiotherapist and on a distal tibiofibular joint of the participant and bulkhead between the limb and the belt, they are placed as two hands of the physiotherapist superimposed non-talus for stabilization. With the posterior removal of the physiotherapist's hip a distal end of the tibia and fibula will be tractioned and maintained anteriorly, while requested that the participant performed an active knee flexion movement in a closed kinetic chain in order to force the movement of ankle dorsiflexion And thus, once the end point for the purpose, a mobilization will be held for 10 seconds. The patient will return to the starting point resting for 20 seconds for a next mobilization. In all, 4 separate mobilizations.

Placebo intervention: The positioning of the hand in the specific treatment condition (Thrust or MWM) will be accurately reproduced, however, without any movement or force being applied. All interactions, procedures and deadlines are identical.

ELIGIBILITY:
Inclusion Criteria:

* Be a regular practitioner of some sporting modality (with a minimum of one year of practice and training frequency of twice a week), with a history of at least one unilateral ankle sprain with episodes of pain and decreased function, as well as a subjective report of Ankle instability (sensation of falsehood) after ligament injury associated with a result lower than 24 points in the Portuguese version of the Cumberland Ankle Instability Tool - CAIT

Exclusion Criteria:

* Participants with acute or subacute lesions and / or lower limb surgery.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-01-30 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Balance assessed with Biodex Balance System | almost 10 minutes
  Balance assessed with Biodex Balance System (stabilometry plattaform)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Lima, PhD, Principal Investigator — UFC - DEFISIO
Locations (1):
- Universidade Federal do Ceará, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No